CLINICAL TRIAL: NCT04775368
Title: Syndrome Fibromyalgique en France : Place de l'évaluation et de la Prise en Charge Des Troubles du Sommeil
Brief Title: Fibromyalgia Syndrome in France: The Role of Assessment and Management of Sleep Disorders
Acronym: FIBOBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Emile Roux (Other)
Collaborators: Walisco (Unknown); University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: RIPH2_ANDRE_FIBOBS; 2020-A02940-39 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2021-02-23; First posted 2021-03-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnosis orientation group (Experimental): For this study, there is only one arm. Each patient complete diagnosis questionnaires.
  Interventions: Other: Administering diagnosis orientation questionnaires for the screening of possible sleep disorders

INTERVENTIONS:
Other: Administering diagnosis orientation questionnaires for the screening of possible sleep disorders — Several diagnosis orientation self-questionnaires will be conducted by the patient following his or her inclusion in order to detect, among other things, possible sleep disorders.

SUMMARY:
The FIBOBS study is a multi-centered, observational, prospective study carried out within specialized chronic pain structures (CPS) in France. It will estimate the prevalence of sleep disorders, divided into three categories (poor quality of sleep in general, sleep apnea syndrome, restless legs syndrome), using self-questionnaires in patients with Fibromyalgia Syndrome (FMS) consulting within a CPS. The interaction between these sleep disorders and other symptoms of FMS will also be analyzed using self-administered questionnaires. Based on the hypothesis that sleep disorders associated with FMS are only imperfectly assessed and/or treated in CPS, the FIBOBS study will also interview pain physician in order to know both the diagnostic tools used and the recommended management when sleep disorders are suspected in the context of FMS. In addition, this study will provide a better understanding of the symptoms of FMS, their impact and how patients feel.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Read, write and understand the French language
* Patient with a diagnosis of Fibromyalgia Syndrome according to ACR 2010 criteria: Painful symptoms present at the same intensity for at least 3 months, WPI ≥ 7 and SSS ≥ 5 OR 3 ≤ WPI ≤ 6 and SSS ≥ 9, Any other cause responsible for chronic osteoarticular pain must be excluded.Primary or secondary fibromyalgia is eligible, at the discretion of the investigator.
* Patient seen in consultation for the first time or for a follow-up visit if the patient has already been followed up in the specialized chronic pain structure for less than a year.
* Have access to an internet connection (for the realization of the "patient questionnaire")
* Patient affiliated to a social security system
* Written and signed informed consent

Exclusion Criteria:

* Patient undergoing anti-cancer treatment or having completed treatment less than 2 years ago
* Patient under guardianship, deprived of liberty, safeguard of justice
* Pregnant or breastfeeding women
* Patient presenting a serious psychiatric pathology that does not allow compliance with the completion of the questionnaires (at the discretion of the investigator)
* Refusal to participate in research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 601 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
Assessing the prevalence of sleep disorders in general in patients with FMS | Only once, by the patient within 14 days of inclusion.
  The prevalence of sleep disorders will be estimated from the results of the Pittsburgh Sleep Quality Index Questionnaire (PSQI) which is a generic, validated 19-item self-administered questionnaire for measuring sleep problems.
Assessing the prevalence of sleep disorders for the specific risk of sleep apnea syndrome in patients with FMS | Only once, by the patient within 14 days of inclusion.
  The prevalence of sleep disorders for the specific risk of sleep apnea syndrome will be estimated from the results of the STOP-BANG questionnaire. This questionnaire guide the diagnosis of sleep apnea syndrome and is composed of 8 items.
Assessing the prevalence of sleep disorders for the specific risk of restless legs syndrome in patients with FMS | Only once, by the patient within 14 days of inclusion.
  The prevalence of sleep disorders will be estimated from the results of the simple question which is a rapid screening tool that provides a diagnosis of probable restless legs syndrome (RLS). Patients who answer positively to this question will complete the International Restless Legs Syndrome (IRLS) questionnaire which assesses the severity of restless legs syndrome on four levels: mild, moderate, severe and very severe.

SECONDARY OUTCOMES:
Assessing the pain severity of FMS | Only once, by the patient within 14 days of inclusion.
  The pain severity of the FMS will be assessed using the WPI (widespread pain index) questionnaire, which represents the generalized pain index.
Assessing the symptom severity of FMS | Only once, by the patient within 14 days of inclusion.
  The symptom severity of the FMS will be assessed using the SSS (symptom severity scale) questionnaire, which corresponds to the symptom severity scale.
Assessing the impact of the FMS on the patient's daily life | Only once, by the patient within 14 days of inclusion.
  The impact of the FMS on the patient's daily life will be assessed by the QIF (French version of the Fibromyalgia Impact Questionnaire (FIQ)). This validated and commonly used questionnaire makes it possible to evaluate the functional incapacity and the repercussions of the FMS on daily life by evaluating the major symptoms: pain, fatigue, sleep disorders but also morning stiffness, anxiety and depression.
Assessing the feeling of pain and the impact of pain on the patient's daily behavior | Only once, by the patient within 14 days of inclusion.
  The painful feeling and the impact of pain on the patient's daily behavior will be assessed by the Concise Pain Questionnaire (QCD), the French version of the Brief Pain Inventory (BPI). This validated questionnaire makes it possible to assess the impact of pain on seven general aspects of the patient's life.
Assess the patient's state of anxiety and depression | Only once, by the patient within 14 days of inclusion.
  The patient's state of anxiety and depression will be assessed using the validated HADS - Hospital Anxiety and Depression Scale questionnaire.
Describe the assessment tools used by the pain physician to evaluate the main symptoms of FMS (pain, asthenia, sleep and cognitive disorders) | Only once, by the pain physician at the inclusion.
  The assessment tools used by the pain physician to evaluate patients' pain, asthenia, sleep disorders and memory problems will be recorded in the "physician questionnaire".
Describe the therapeutic measures (drug and non-drug) in place for the management of FMS | Once by the physician at the inclusion, and once by the patient within 14 days of inclusion.
  Therapeutics proposed for the management of symptoms associated with FMS will be identified (names of drug and non-drug treatments, care practices).
Assess the percentage of patients for whom sleep disorders have been previously diagnosed and treated. | Throught study completion, an average of 4 months.
  The "patient questionnaire" will identify patients already diagnosed and treated for a sleep disorder. This will allow comparison with the prevalence calculated from the three screening questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert ANDRE, MD, Principal Investigator — CH Emile Roux - Le Puy-en-Velay
Locations (46):
- France (46):
  - CHU Amiens Picardie - CETD, Amiens
  - CH Ardèche Méridionale, Aubenas
  - CH Henri Mondor, Aurillac
  - CHU Jean Minjoz - CETD, Besançon
  - CH Béziers, Béziers
  - HIA Clermont Tonnerre, Brest
  - CHU Hôpital Côte de Nacre - CETD, Caen
  - CH Métropole Savoie, Chambéry
  - CH de Chartres, Chartres
  - CHU Gabriel Montpied, Clermont-Ferrand
  - CH du Pays de Craponne, Craponne-sur-Arzon
  - CH de Dax, Dax
  - Centre Hospitalier de Dieppe, Dieppe
  - CH de Dreux, Dreux
  - CHI Fréjus - Saint Raphaël, Fréjus
  - GMH, Grenoble
  - CHD Vendée, La Roche-sur-Yon
  - GH Littoral Atlantique, La Rochelle
  - CHU Grenoble Alpes, La Tronche
  - CH Pierre Gallice, Langeac
  - CH de Versailles, Le Chesnay
  - Centre Hospitalier du Mans, Le Mans
  - CH Emile Roux, Le Puy-en-Velay
  - CHU Dupuytren 2 - Centre de la douleur chronique, Limoges
  - Clinique Mutualiste de la Porte de Lorient, Lorient
  - Centre de la douleur Lille métropole, Marquette-lez-Lille
  - CHU Timone, Marseille
  - Hôpital Sainte Blandine, Metz
  - CHI de Mont-de-Marsan, Mont-de-Marsan
  - CH du Forez, Montbrison
  - GHR MSA - CETD - Site Muller, Mulhouse
  - CHU Nord, Nantes
  - CHR Orléans, Orléans
  - GH Paris Saint Joseph, Paris
  - CH de Perpignan, Perpignan
  - CHU de Poitiers, Poitiers
  - CH René Dubos, Pontoise
  - CH Annecy Genevois, Pringy
  - CHU de Saint-Etienne, Saint-Etienne
  - CH Saint-Nazaire, Saint-Nazaire
  - Hôpital Pierre Paul Riquet - CHU Toulouse, Toulouse
  - CH de Valence, Valence
  - CH Jacques Lacarin, Vichy
  - Hôpital Nord Ouest - Site Villefranche-sur-Saône, Villefranche-sur-Saône
  - Médipôle Hôpital Mutualiste, Villeurbanne
  - CH Jacques Barrot, Yssingeaux

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andre G, Petitjean P, Haas V, Geraud E, Fantini ML, Creac'h C, Perez C, Bonnefoi M, Gadea E. Screening and management of sleep disorders in patients with fibromyalgia syndrome: a French multicentred, prospective, observational study protocol (FIBOBS). BMJ Open. 2022 Sep 30;12(9):e062549. doi: 10.1136/bmjopen-2022-062549. PMID 36180114